CLINICAL TRIAL: NCT04746976
Title: A Prospective, Observational Study Evaluating Persistence on Treatment, Safety, Tolerability, and Effectiveness of Diroximel Fumarate in the Real-World Setting (EXPERIENCE-US Study)
Brief Title: Study of Diroximel Fumarate in the Real-World Setting
Status: Terminated | Type: Observational
Why Stopped: Sponsor's Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-VUM-11760
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Relapsing Forms of MS
Keywords: Clinically isolated syndrome; Multiple Sclerosis; Relapsing forms of Multiple Sclerosis; Active secondary progressive disease
MeSH Terms: conditions — Multiple Sclerosis | interventions — diroximel fumarate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diroximel Fumarate: Participants with RMS who are receiving diroximel fumarate orally in routine clinical practice will be enrolled.
  Interventions: Drug: Diroximel Fumarate

INTERVENTIONS:
Drug: Diroximel Fumarate — As described in the arm.
  Other Names: VUMERITY; BIIB098

SUMMARY:
The primary objective of the study is to characterize the persistence to therapy in participants with relapsing forms of multiple sclerosis (RMS) treated with diroximel fumarate (DRF) in routine clinical practice. The secondary objectives of the study are to assess short-term persistence to treatment; to assess long-term persistence on treatment; to assess the effect of DRF on relapses; to assess the impact of DRF on cognition; to assess the impact of DRF on participant reported outcomes (PROs) and to explore the real-world safety profile of DRF (ie, gastrointestinal [GI] tolerability, lymphocyte dynamics, adverse events [AEs] leading to discontinuation, and serious adverse events [SAEs]).

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of MS and satisfy the approved therapeutic indication for DRF per the USPI.
* DRF prescribed and planned to be initiated within 60 days after enrollment.

Key Exclusion Criteria:

* History of gastric bypass or required use of feeding tubes.
* Have received prior treatment with DRF.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with Relapsing forms of multiple sclerosis (RMS) that have been prescribed Diroximel Fumarate under standard clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants on Treatment with DRF at 1 Year | 1 year

SECONDARY OUTCOMES:
Percentage of Participants on Treatment with DRF at 3 Months | 3 months
Percentage of Participants on Treatment with DRF at 2 Years | 2 years
Annualized Relapse Rate (ARR) with DRF | At 1 and 2 years
Percentage of Participants Relapsed | At 1 and 2 years
Change in Processing Speed Test (PST) Score from Baseline | Baseline up to 2 years
  PST measures mental processing speed. The PST will be assessed using multiple sclerosis performance test (MSPT). The participants will be shown some symbols and corresponding numbers. The participants will be then asked to input the numbers corresponding to the given symbols in empty rows. Higher number of correct responses indicates better cognition
Change in Score for Each Domain of Quality of Life in Neurological Disorders (Neuro- QoL™) Questionnaire | Baseline up to 2 years
  Neuro-QOL uses a T score which has a mean of 50 and SD of 10, based on the norming sample used. All Neuro-QOL banks and scales are scored such that a high score reflects more of what is being measured.
Change in Disability, as Measured by Patient Determined Disease Steps (PDDS) | Baseline up to 2 years
  The PDDS has nine ordinal levels ranging between 0 (normal) and 8 (bedridden). Higher scores indicate greater disability.
Change in Work Productivity and Activity Impairment Due to Multiple Sclerosis (WPAI- MS) Scores from Baseline | Baseline up to 2 years
  The Work Productivity and Activity Impairment (WPAI) questionnaire is a validated instrument to measure impairments in work and activities. The WPAI yields four types of scores: 1. Absenteeism (work time missed) 2. Presenteesism (impairment at work / reduced on-the-job effectiveness) 3. Work productivity loss (overall work impairment / absenteeism plus presenteeism) 4. Activity Impairment. Higher numbers indicate greater impairment and less productivity.
Number of Participants with Gastrointestinal (GI) Adverse Events (AEs) | Up to 32 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with AEs Leading to Treatment Discontinuation | Up to 32 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal assessment such as an abnormal laboratory value), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Number of Participants with Serious Adverse Events (SAEs) | Up to 32 months
  An SAE is any untoward medical occurrence that at any dose results in death, in the view of the investigator, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.
Number of Participants categorized by the types of actions taken to mitigate GI AEs | Up to 32 months
  The actions taken will include temporary dose reduction, temporary dose interruption, initiation of concomitant GI medication, taking DRF dose with food, permanent discontinuation, or other action.
Median Absolute Lymphocyte Count (ALC) Over Time | Baseline up to 2 years
Percent Change in Median ALC from Baseline | Baseline up to 2 years
Number of Participants with Lymphopenia According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI/CTCAE)Severity Grading | Up to 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (18):
- United States (18):
  - Regina Berkovich MD Phd Inc, West Hollywood, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Norton Neuroscience Institute, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Glendale Neurological Associates, PC, Farmington, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - St. Luke's Neurology, Kansas City, Missouri
  - CentraState Healthcare System - Linda Cardinale MS Center, Freehold, New Jersey
  - MS Center at St Barnabas, Livingston, New Jersey
  - Multiple Sclerosis Center JSUMC, Neptune City, New Jersey
  - Jacobs School of Medicine and Biomedical Sciences, Buffalo, New York
  - Cone Health, Greensboro, North Carolina
  - Providence Brain and Spine Institute, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Hope Neurology, Knoxville, Tennessee
  - UTHealth Neurosciences Texas Medical Center II, Houston, Texas
  - Riverside Neurology Specialists, Newport News, Virginia
  - Providence Medical Research Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/